CLINICAL TRIAL: NCT05691829
Title: A Phase II Trial of Immunotherapy With Non-Ablative Radiation in Previously Untreated Patients With Stage IV NSCLC
Brief Title: Immunotherapy With Non-Ablative Radiation in Previously Untreated Patients With Stage IV NSCLC
Acronym: IRRADIATE-Lung
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to insufficient enrollment.
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-00673
Record Dates: First submitted 2023-01-11; First posted 2023-01-20 (Actual); Results first posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: NSCLC Stage IV
Keywords: Lung; Immunotherapy; Fraction non-ablative radiation; untreated patients; metastatic
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis | interventions — pembrolizumab; Radiation; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Untreated Patients With Stage IV NSCLC (Experimental): Participants will receive radiation in concert with starting chemotherapy with pembrolizumab for up to 6 cycles (18 weeks), followed by continued treatment with pembrolizumab (standard of care). Patients will be followed for 1 year following the completion of the core study period of 6 cycles.
  Interventions: Drug: Pembrolizumab; Radiation: Radiation; Drug: Chemotherapy

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab 200mg solution administered intravenously every 3 weeks for 6 cycles followed by maintenance therapy until progression of disease or unacceptable toxicity (standard of care). Administered alongside chemotherapy.
  Other Names: MK-3475
Radiation: Radiation — One-time, up-front radiation delivered at up to five metastatic subsites at a 4 Gy x 5 radiation dose fractionation schedule. Radiation will be delivered within five days before or after initiation of first cycle of pembrolizumab treatment. Radiation modality and technique will be determined at the discretion of the treating radiation oncologist.
Drug: Chemotherapy — Administered alongside pembrolizumab every 3 weeks for 6 cycles per institutional standard of care. For non-squamous, the standard chemotherapy option of choice is carboplatin and pemetrexed. For squamous cell carcinoma, the chemotherapy used would be carboplatin and paclitaxel or nab-paclitaxel

SUMMARY:
The purpose of this study is to test if low dose radiation, which is routinely used in treating patients with lung cancer for symptom control, can improve the results from the standard treatment with pembrolizumab and chemotherapy. In this study, only individuals who have NSCLC that is advanced (Stage IV), or has come back (recurred), will be able to participate.

DETAILED DESCRIPTION:
This is a phase II open-label trial of pembrolizumab sequentially following upfront non-ablative focal therapy to up to five distinct metastatic subsites in de novo stage IV Non-Small Cell Lung Cancer (NSCLC). The primary goal of this trial is to evaluate the efficacy defined by time to progression or death with upfront non-ablative focal radiation (RT) to index lesions as a way of enhancing the anti-tumor immune response to pembrolizumab. Adult patients with metastatic NSCLC, with at least 2 measurable lesions and those Patients with metastatic NSCLC who are previously untreated are eligible for the study if they meet all inclusion criteria, and do not satisfy any exclusion criteria. Participants will receive standard of care immunotherapy of Pembrolizumab in addition to non-ablative radiation. The intervention is the low dose fractionation, 4Gy x 5, in the upfront treatment of de novo stage IV NSCLC in up to five distinct subsites of metastatic NSCLC.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent/assent for the trial.
2. Histologically documented, metastatic NSCLC with no previous systemic therapy
3. At least 2 distinct measurable metastatic sites, which are 1 cm or larger; patients can have radiation to multiple measurable disease sites as clinically indicated, however, there must be at least 1 measurable non-radiated target lesion for response assessment.
4. Agreeable to provide archival tissue for correlative studies; if no archival tissue available may obtain an exemption by the study team.
5. Be at least 18 years of age on day of signing informed consent.
6. Have measurable disease based on RECIST 1.1.
7. Have a performance status of ≤1 ECOG Performance Scale.
8. Demonstrate adequate organ function as defined in Table 2, all screening labs should be performed within 10 days of treatment initiation
9. Have one measurable lesion of at least 1 cm outside the planned radiation field (defined as not receiving direct beam from any of the treatment portals).
10. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
11. Female subjects of childbearing potential must be willing to use an adequate method of contraception as outlined in Section - Contraception, for the course of the study through 120 days after the last dose of study medication. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
12. Male subjects of childbearing potential must agree to use an adequate method of contraception as outlined in Section- Contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

Exclusion Criteria:

1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
2. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
3. Has a known history of active TB (Bacillus Tuberculosis)
4. Hypersensitivity to pembrolizumab or any of its excipients.
5. Has had prior chemotherapy, immunotherapy or targeted small molecule therapy within 6 months prior to study Day 1.
6. Patient who have previously received radiation overlapping, as determined by the treating radiation oncologist, with the current planned radiation treatment fields are ineligible.
7. Patient's treated with whole brain radiation therapy are ineligible.
8. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
9. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases (with SRS and/or neurosurgery) may participate provided they are clinically stable and, have no evidence of new or enlarging brain metastases and also are off steroids 3 days prior to dosing with study medication.
10. Patients who have not recovered (i.e., ≤ Grade 2 or at baseline) from adverse events due to a previously administered agent. *Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
11. Has history of autoimmune disorders, (non-infectious) pneumonitis that required steroids, evidence of interstitial lung disease or active, non-infectious pneumonitis.
12. Has an active infection requiring systemic therapy.
13. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
14. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
15. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
16. Patients with prior history of chemoradiation for lung cancer
17. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
18. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
19. Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however, intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2023-01-24 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2025-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vamsidhar Velcheti, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: Vamsidhar.Velcheti@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to Vamsidhar.Velcheti@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Untreated Patients With Stage IV NSCLC
Started | 19
Completed | 14
Not Completed | 5
Not completed — Physician Decision | 2
Not completed — Eligibility criteria not met | 3

BASELINE CHARACTERISTICS:
Arm/Group | Untreated Patients With Stage IV NSCLC
Number analyzed (Participants) | 14
Age, Continuous [Median (Full Range); unit: years] | 80 [46 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 8
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants With a Best Overall Response of Complete Response (CR) or Partial Response (PR) by End of Treatment Cycle 4
Description: Defined as the best response recorded from the start of the study treatment until the end of treatment Cycle 4, either Complete Response or Partial Response. A CR is defined as the disappearance of all target lesions (TLs) and reduction in the short axis measurement of all pathologic lymph nodes to ≤10 mm. A PR is defined as at least a 30% decrease in the sum of the longest diameter (SLD) of TLs, taking as reference the baseline SLD.
Time Frame: Up to Week 12 (End of Cycle 4 - each cycle is 21 days)
Population: 1 participant did not start treatment
Measure: Number; unit: percentage of participants
Arm/Group | Untreated Patients With Stage IV NSCLC
Number analyzed (Participants) | 13
percentage of participants | 30.77

2. Secondary Outcome: Progression-Free Survival (PFS) at Final Follow-Up
Description: PFS is defined as the time from initiation of study drug post-radiation, until the first documented, confirmed progression of disease or death.
Time Frame: From enrollment until the first documented and confirmed progression of disease, death, date last follow-up, or end of study; assessed up to 81 weeks
Population: 1 participant did not start treatment
Measure: Median (Full Range); unit: weeks
Arm/Group | Untreated Patients With Stage IV NSCLC
Number analyzed (Participants) | 13
weeks | 42.86 [6.43 to 80.86]

3. Secondary Outcome: Overall Survival (OS) at Final Follow-Up
Description: OS is defined as the time (in weeks) to death from the start of drug therapy.
Time Frame: as for outcome 2
Population: 1 participant did not start treatment
Measure: Median (Full Range); unit: weeks
Arm/Group | Untreated Patients With Stage IV NSCLC
Number analyzed (Participants) | 13
weeks | 51.57 [6.43 to 80.86]

4. Secondary Outcome: Percentage of Participants With an Objective Response
Description: An objective response (Complete Response or Partial Response) is defined as lasting continuously for 6 months and starting any time within 12 months of initiating therapy. A CR is defined as the disappearance of all target lesions and reduction in the short axis measurement of all pathologic lymph nodes to ≤10 mm. A PR is defined as at least a 30% decrease in the sum of the longest diameter (SLD) of TLs, taking as reference the baseline SLD.
Time Frame: Week 52
Population: 1 participant did not start treatment
Measure: Number; unit: percentage of participants
Arm/Group | Untreated Patients With Stage IV NSCLC
Number analyzed (Participants) | 13
percentage of participants | 38.46

ADVERSE EVENTS:
Time Frame: AE monitoring: from time of consent through 30 days post treatment (up to 22 weeks) All cause mortality monitoring: from time of consent until End of Study (up to 81 weeks)
Description: Investigators reviewed adverse events at every study visit (every 3 weeks).
Arm/Group | Untreated Patients With Stage IV NSCLC
All-Cause Mortality (participants affected / at risk) | 4/14
Serious Adverse Events (participants affected / at risk) | 9/14
Other Adverse Events (participants affected / at risk) | 13/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Untreated Patients With Stage IV NSCLC (N=14)
Abdominal Pain (Gastrointestinal disorders) | 1
Adrenal Insufficiency (Nervous system disorders) | 1
Arterial Thomboembolism (Vascular disorders) | 1
Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 1
Disease Progression (General disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Heart Failure (Cardiac disorders) | 1
Injury, Other (Injury, poisoning and procedural complications) | 1
Intracranial Hemorrhage (Nervous system disorders) | 1
Lung Infection: Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Massive Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Multiple Fractures From Trauma (Injury, poisoning and procedural complications) | 1
Urinary Tract Infection (Renal and urinary disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Untreated Patients With Stage IV NSCLC (N=14)
Skin, Other: Wounds From Trauma (Skin and subcutaneous tissue disorders) | 1
ANC Decreased (Blood and lymphatic system disorders) | 2
Anemia (Blood and lymphatic system disorders) | 2
Anorexia (Metabolism and nutrition disorders) | 2
Appetite (Metabolism and nutrition disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 2
Chest Pain, Non-Cardiac (Respiratory, thoracic and mediastinal disorders) | 1
Chest Wall Pain (Non-Cardiac: ribcage) (Respiratory, thoracic and mediastinal disorders) | 1
Constipation (Gastrointestinal disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Covid 19 Virus (Respiratory, thoracic and mediastinal disorders) | 2
Creatinine Increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Dry Mouth (Gastrointestinal disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Edema Limbs (General disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Erythematous Rash (Skin and subcutaneous tissue disorders) | 1
Fatigue (General disorders) | 5
Fever (General disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Herpes Simplex Virus (Infections and infestations) | 1
Hoarseness (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Hypotension (Vascular disorders) | 1
Insomnia (Psychiatric disorders) | 3
Intermittent Diarrhea (Gastrointestinal disorders) | 1
Intermittent Nausea (Gastrointestinal disorders) | 1
Knee Pain / Gout (Musculoskeletal and connective tissue disorders) | 1
Left Arm Paresthesia (Nervous system disorders) | 1
Lower Extremity Muscle Cramps (Musculoskeletal and connective tissue disorders) | 1
Lower Extremity Weakness (Musculoskeletal and connective tissue disorders) | 1
Lymphocyte Count Decreased (Investigations) | 4
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Oral Dysesthesia (Gastrointestinal disorders) | 1
Other Respiratory Symptom (Respiratory, thoracic and mediastinal disorders) | 1
Pain (Groin, Right-Sided, Post-Operative) (Injury, poisoning and procedural complications) | 1
Pain (Multiple Bone Fractures) (Injury, poisoning and procedural complications) | 1
Pain In Extremity (B/L Back Thighs) (Musculoskeletal and connective tissue disorders) | 1
Pain, R Foot (Musculoskeletal and connective tissue disorders) | 1
Palmar (Skin and subcutaneous tissue disorders) | 1
Papulopustular Rash (Skin and subcutaneous tissue disorders) | 1
Paresthesia (Right Foot) (Nervous system disorders) | 1
Periorbital Edema (Eye disorders) | 1
Peripheral Neuropathy (Nervous system disorders) | 1
Platelet Count Decreased (Investigations) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3
Purulent Tear Discharge (Eye disorders) | 1
Rash On Leg (Skin and subcutaneous tissue disorders) | 1
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 2
Sinus Tachycardia (Cardiac disorders) | 1
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 2
Tachycardia (Cardiac disorders) | 1
Thrombolic Event (Vascular disorders) | 1
Urinary Frequency (Renal and urinary disorders) | 1
Urinary Retention (Renal and urinary disorders) | 1
Vaginal Infection (Infections and infestations) | 1
WBC Decreased (Investigations) | 2
Weight Loss (Investigations) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-09): https://cdn.clinicaltrials.gov/large-docs/29/NCT05691829/Prot_SAP_000.pdf